CLINICAL TRIAL: NCT01891682
Title: Methionine Metabolism in Parenterally Fed Critically Ill Children
Brief Title: Methionine Metabolism in Parenterally Fed Pediatric Sepsis
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Leticia Castillo, Department Chair Peds Critical Care, The Cleveland Clinic
Other Study IDs: STU-022012-035
Record Dates: First submitted 2013-06-24; First posted 2013-07-03 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Sepsis; Critical Illness
Keywords: Methionine Metabolism; Parenteral Nutrition; Pediatric; Pediatrics; Sepsis; Observational Study
MeSH Terms: conditions — Sepsis; Critical Illness; Hyperphagia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Critically Ill Pediatric Patients: Critically ill septic pediatric patients, Age 1 month-3 years, Age 4-12 years and Age 13-19 years, males and females
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational, Translational non-treatment study

SUMMARY:
Critically ill children have abnormal utilization of nutrients such as glucose, lipids and protein. Protein synthesis is increased mainly in the form of immune and signaling proteins, while synthesis of muscle and structural proteins is decreased. The metabolism of sulfur amino acids and specifically methionine and cysteine have not been investigated in critically ill septic children, despite that sulfur amino acids have important roles on thiol, antioxidant and epigenetic reactions, as well as precursor of glutathione (GSH). Methionine metabolism in critically ill children will be influenced by its rate of utilization through the transmethylation, remethylation and transsulfuration pathways, which are the major pathways of methionine metabolism.

The investigators study aims to investigate the metabolism of methionine and cysteine in parenterally fed critically ill septic children. The investigators aim to determine the rates of transmethylation, remethylation, transsulfuration and GSH synthesis rates in critically ill septic children, to determine in vivo, whole body sulfur amino acid metabolism when sulfur amino acids are supplied by the parenteral route. The objective is to determine whether current parenteral intakes support GSH synthesis and if methionine metabolism differs when supplied by the parenteral versus the enteral route. Methionine parenteral requirements will be also studied by using the indicator amino acid oxidation and balance technique.

DETAILED DESCRIPTION:
This is a prospective, translational study on whole body methionine metabolism and requirements when administered by the parenteral route in critically ill septic children. The study size will include 45 critically ill septic, pediatric patients (15 infants at 1 month-3 years of age, 15 children at 4-12 years of age and 15 adolescent at 13-19 years of age, male and females admitted to the pediatric intensive care unit (PICU) at Children's Medical Center, Dallas. The minimal subject's weight will be 4 kg. The number of subjects includes an expected drop out rate of about 20%, in order to obtain 12 patients with complete data in each group. Patients will receive nutritional support as per standard care. This study will yield important knowledge and may lead in the future to changes in the current practice on the management of critically ill pediatric patients in the PICU.

Study Aim#1: Determine the parenteral requirements of methionine, in the presence of cysteine, in critically ill septic patients' required extended use of TPN, by using the indicator amino acid oxidation and balance technique.

Study Aim#2: Determine methionine metabolism through the rates of transmethylation, transsulfuration and remethylation at the current standard intakes of methionine of 120 mg.kg.d. with negligible amounts of cysteine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 month-19 years
2. Diagnosis of severe sepsis diagnosed as clinical sepsis syndrome (requires two of the following criteria):

   * Source of infection
   * Fever or Hypothermia
   * Leukocytosis or Leucopenia
   * Poor organ perfusion (such as delayed capillary refill or decreased urine output or hypotension)
   * Bacteremic sepsis demonstrated by positive blood culture
3. Weight greater or equal to 4 kg
4. Need for parenteral nutrition
5. Presence of central and/or arterial venous access as per clinical indication

Exclusion Criteria:

1. Patients with metabolic diseases (i.e. Insulin dependent diabetes mellitus, urea cycle disorders, cystinuria, etc.)
2. Pregnancy
3. Primary liver failure
4. Primary renal failure
5. Patients on enteral feedings greater than 20% of daily requirement
6. Weight less than 4.0 kg

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Septic pediatric patients: A total of 45 critically ill children age 1 month-19 years with diagnosis of sepsis, as defined by the International Sepsis Consensus Conference.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Parenteral Requirements of Methionine | 8 hours
  Breakpoint between the rates of indicator amino acid oxidation and level of parenteral methionine intake.

SECONDARY OUTCOMES:
Methionine Metabolism | 8 hours
  Rates of transmethylation, remethylation and transsulfuration and erythrocyte GSH synthesis when nutrients are given by the parenteral route in pediatric critically ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Castillo, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States